CLINICAL TRIAL: NCT05359575
Title: Measuring the Effectiveness of Three Instructional Interventions for Prehospital Cervical Spinal Immobilization by Laypeople: A Randomized Clinical Trial
Brief Title: Three Instructional Interventions for Prehospital Cervical Spinal Immobilization by Laypeople
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Washington University School of Medicine (Other); LFR International (Unknown)
Responsible Party: Principal Investigator, Jaimo Ahn, Harold W. and Helen L. Gehring Research Professor of Orthopedic Surgery, University of Michigan
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: HUM00210308
Record Dates: First submitted 2022-04-23; First posted 2022-05-04 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: Cervical Vertebra Injury; Cervical Vertebra Fracture

STUDY DESIGN:
Intervention Model Description: Participants are initially randomized to 1 of 4 arms. Once the initial instructional intervention is completed, participants are subsequently randomized to either a 1-month or 2-month follow-up.
  Participants initially randomized to the two arms with flashcards (v. 1) are not randomized to either follow up, because version 1 of the flash cards was confusing and thus was piloted with these initial participants.
Who Masked: Outcomes Assessor
Masking Description: The outcomes assessor only enters the laboratory after the participant has attempted to apply the cervical collar (c-collar). Therefore, the outcomes assessor is unaware of the instructional intervention that was employed. The outcomes assessor will collect cervical range of motion (CROM) measurements using a CROM device to verify correct c-collar placement by evaluating whether the c-collar was appropriately sized and if neck movement is restricted in five cardinal directions: flexion, extension, and bidirectional rotation.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (10):
- Audio recording with instructional flashcard with cervical-collar ("audio kit") - 1 month follow-up (Experimental): MP3 audio files for each of 6 steps (totaling 1 minute, 19 seconds) and instructional flashcard with seven pictures corresponding to each of the 6 steps of c-collar application, used for c-collar application attempt. Participants repeat the c-collar application with the audio kit at 1 month follow-up.
  Interventions: Behavioral: Audio kit; Behavioral: Instructional flashcard (version 2)
- Instructional flashcard with cervical-collar - 1 month follow-up (Experimental): Instructional flashcard with seven pictures corresponding to 6 steps of c-collar application, used for c-collar application attempt. Participants repeat the c-collar application with the instructional flashcard at 1 month follow-up.
  Interventions: Behavioral: Instructional flashcard (version 2)
- In-person training with cervical-collar - 1 month follow-up (Experimental): 10 minutes of a Lay First Responder (LFR) spinal immobilization course (extracted from the current LFR Level 1 trauma course) are used for instruction for c-collar application attempt. Participants repeat the c-collar application without any POC instruction or re-training at 1 month follow-up.
  Interventions: Behavioral: In-person training
- Control group with no in-person training and no access to POC instruction - 1 month follow-up (No Intervention): There is no in-person training or point-of-care (POC) instructional interventions for this group for c-collar application attempt. Participants repeat the c-collar application without any in-person training or POC instructional interventions at 1 month follow-up.
- Audio recording with instructional flashcard with cervical-collar ("audio kit") - 2 Months follow-up (Experimental): MP3 audio files for each of 6 steps (totaling 1 minute, 19 seconds) and instructional flashcard with seven pictures corresponding to each of the 6 steps of c-collar application, used for c-collar application attempt. Participants repeat the c-collar application with the audio kit at 2 months follow-up.
  Interventions: Behavioral: Audio kit; Behavioral: Instructional flashcard (version 2)
- Instructional flashcard with cervical-collar - 2 months follow-up (Experimental): Instructional flashcard with seven pictures corresponding to 6 steps of c-collar application, used for c-collar application attempt. Participants repeat the c-collar application with the instructional flashcard at 2 months follow-up.
  Interventions: Behavioral: Instructional flashcard (version 2)
- In-person training with cervical-collar - 2 months follow-up (Experimental): 10 minutes of a Lay First Responder (LFR) spinal immobilization course (extracted from the current LFR Level 1 trauma course) are used for instruction for c-collar application attempt. Participants repeat the c-collar application without any POC instruction or re-training at 2 months follow-up.
  Interventions: Behavioral: In-person training
- Control group with no in-person training and no access to POC instruction - 2 months follow-up (No Intervention): There is no in-person training or POC instructional interventions for this group for c-collar application attempt. Participants repeat the c-collar application without any in-person training or POC instructional interventions at 2 months follow-up.
- Audio recording with instructional flashcard (version 1) with cervical-collar - no follow-up (Experimental): Prior to randomization to 1 or 2 month follow up, these participants served as an initial cohort of participants who were not assigned to any longitudinal follow-up date so that the POC instructional flashcard could first be piloted to receive feedback for instructional flashcard revision prior to launching the "trial" after participants expressed concern about ambiguity in the instructional flashcard. Data from these participants is not considered part of the "trial" for any analytic purposes. Revisions to the instructional flashcard were made.
  Interventions: Behavioral: Audio kit; Behavioral: Instructional flashcard (version 1)
- Instructional flashcard (version 1) with cervical-collar - no follow-up (Experimental): Prior to randomization to 1 or 2 month follow up, these participants served as an initial cohort of participants who were not assigned to any longitudinal follow-up date so that the POC instructional flashcard could first be piloted to receive feedback for instructional flashcard revision prior to launching the "trial" after participants expressed concern about ambiguity in the instructional flashcard. Data from these participants is not considered part of the "trial" for any analytic purposes. Revisions to the instructional flashcard were made.
  Interventions: Behavioral: Instructional flashcard (version 1)

INTERVENTIONS:
Behavioral: Audio kit — MP3 audio files for each of 6 steps of c-collar application (totaling 1 minute, 19 seconds) and instructional flashcard with seven pictures corresponding to each of the 6 steps of c-collar application
  Arms: Audio recording with instructional flashcard (version 1) with cervical-collar - no follow-up; Audio recording with instructional flashcard with cervical-collar ("audio kit") - 1 month follow-up; Audio recording with instructional flashcard with cervical-collar ("audio kit") - 2 Months follow-up
Behavioral: Instructional flashcard (version 1) — Single page with 7 pictures corresponding to each of the 6 steps of cervical collar (c-collar) application.
  Arms: Audio recording with instructional flashcard (version 1) with cervical-collar - no follow-up; Instructional flashcard (version 1) with cervical-collar - no follow-up
Behavioral: In-person training — 10 minute of an LFR spinal immobilization course (extracted from the current LFR Level 1 trauma course).
  Arms: In-person training with cervical-collar - 1 month follow-up; In-person training with cervical-collar - 2 months follow-up
Behavioral: Instructional flashcard (version 2) — Single page with 7 pictures corresponding to each of the 6 steps of cervical collar (c-collar) application edited for clarity based on initial pilot feedback.
  Arms: Audio recording with instructional flashcard with cervical-collar ("audio kit") - 1 month follow-up; Audio recording with instructional flashcard with cervical-collar ("audio kit") - 2 Months follow-up; Instructional flashcard with cervical-collar - 1 month follow-up; Instructional flashcard with cervical-collar - 2 months follow-up

SUMMARY:
It is not known if bystanders equipped with point-of-care (POC) instruction are as effective as bystanders with in-person training for c-spine immobilization. Therefore, POC instructional interventions were developed during this study in response to the scalability challenges associated with in-person training to measure the comparative effectiveness and skill retention of POC instructions vs in-person training using a randomized clinical trial design.

DETAILED DESCRIPTION:
Road traffic injuries (RTIs) are the largest contributor to the global injury burden, which disproportionately affects low- and middle-income countries (LMICs). Traumatic spinal cord injury (TSCI) is the highest contributor to years lived disabled (YLDs) resulting from RTIs, accounting for 74.8% of YLDs from RTI. With a lack of robust emergency medical services (EMS), there has been increasing reliance on layperson bystanders to respond to RTIs in LMICs. Early spinal immobilization has the potential to limit neurological deficits secondary to TSCI and morbidity. Bystanders may be trained in-person or point-of-care (POC) instruction may be provided, as exists with automated external defibrillators and tourniquets. However, it is unknown if bystanders equipped with POC instruction are as effective as bystanders with in-person training for c-spine immobilization. Therefore, POC instructional interventions were developed in response to the scalability challenges associated with in-person training to measure the comparative effectiveness and skill retention of POC instructions vs in-person training using a randomized clinical trial design. The POC instructional flashcard was first piloted with an initial cohort of participants who were not assigned to any longitudinal follow-up date to pilot POC instructional interventions for c-spine immobilization and receive feedback for instructional flashcard revision prior to launching the "trial." Data from these participants is not considered part of the "trial" for analytic purposes. This entire testing process is with participants who are healthy volunteers and researchers simulating spinal injury victims to test which method of instruction is most effective and durable for understanding.

ELIGIBILITY:
Inclusion Criteria:

* Understand spoken and written English.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 265 (Actual)
Dates: Start 2022-02-07 (Actual); Primary Completion 2022-04-29 (Actual); Study Completion 2022-04-29 (Actual)

PRIMARY OUTCOMES:
Correct c-collar application | After initial intervention (up to 20 minutes)
  Measurement: Number of participants who meet all 4 of the criteria for correct application of the c-collar.
Knowledge retention of correct c-collar application at follow up (1 month) | 1 month
  Measurement: Number of participants who meet all 4 of the criteria for correct application of the c-collar.
Knowledge retention of correct c-collar application at follow up (2 months) | 2 months
  Measurement: Number of participants who meet all 4 of the criteria for correct application of the c-collar.

SECONDARY OUTCOMES:
Level of Participant Confidence | After initial intervention (up to 20 minutes)
  Participants will self-rate on a Likert scale of 0 - 10, where 0 is no confidence and 10 is absolutely confident.
Level of Participant Confidence (1 month) | 1 month
  Participants will self-rate on a Likert scale of 0 - 10, where 0 is no confidence and 10 is absolutely confident.
Level of Participant Confidence (2 months) | 2 month
  Participants will self-rate on a Likert scale of 0 - 10, where 0 is no confidence and 10 is absolutely confident.

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Widder, Study Director — Washington University in St. Louis - McKelvey School of Engineering; Peter Delaney, Study Director — University of Michigan
Locations (1):
- Washington University in St. Louis - McKelvey School of Engineering, Dept. of Biomedical Engineering, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
Upon reasonable request to the corresponding author.
Time Frame: Within 18 months of completion of primary outcome measures.